CLINICAL TRIAL: NCT05644626
Title: A Phase 1a/1b Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-B167, Alone and in Combination With Tislelizumab in Chinese Patients With Selected Advanced or Metastatic Solid Tumors
Brief Title: Safety, Pharmacokinetics and Antitumor Activity of BGB-B167 Alone and in Combination With Tislelizumab in Participants With Solid Tumors in Chinese Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor determined the data was no longer needed.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-B167-102
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1a: Dose Escalation (Experimental): Part A: Increasing dose levels of BGB-B167 monotherapy; Part B: Increasing dose levels of BGB-B167 in combination with tislelizumab (BGB-A317)
  Interventions: Drug: BGB-B167; Drug: Tislelizumab
- Phase 1b: Dose Expansion (Experimental): BGB-B167 alone or in combination with tislelizumab (BGB-A317)
  Interventions: Drug: BGB-B167; Drug: Tislelizumab

INTERVENTIONS:
Drug: BGB-B167 — Intravenous administration
Drug: Tislelizumab — Intravenous administration
  Other Names: BGB-A317

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of BGB-B167 monotherapy and in combination with tislelizumab (BGB-A317) in participants with select advanced solid tumors in Chinese participants

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumors previously treated with standard systemic therapy or for whom treatment is not available, not tolerated, or refused, or not expected to provide significant clinical benefit or be tolerated in the medical judgement of the investigator
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Adequate organ function as indicated by laboratory values during screening or ≤ 7 days before the first dose of study drug(s)
* Women of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study
* Nonsterile men must be willing to use highly effective method of birth control for the duration of the study

Exclusion Criteria:

* Active leptomeningeal disease or uncontrolled, untreated brain metastasis
* Active autoimmune diseases or history of autoimmune diseases that may relapse
* Any malignancy ≤ 3 years before the first dose of study drug(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent
* History of severe hypersensitivity reactions to other monoclonal antibody products or their excipients
* Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers
* Known history of HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Approximately 30 months
Phase 1a: Number of Participants Experiencing AEs Meeting Protocol-defined Dose-limiting Toxicity (DLT) Criteria | Up to Approximately 24 months
Phase 1a: Maximum Tolerated Dose (MTD) of BGB-B167 | Approximately 30 months
  The maximum tolerated dose (MTD) is defined as the highest tolerated dose for which the estimated toxicity rate is closest to the target toxicity rate of 30%.
Phase 1a: Recommended Phase 2 doses (RP2Ds) | Approximately 24 months
  RP2Ds of BGB-B167 alone or in combination with tislelizumab will be determined based on a biologically effective dose
Phase 1b: Objective Response Rate (ORR) as determined by investigators per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to Approximately 30 months
  ORR is defined as the proportion of participants who had confirmed complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Phase 1a: ORR | Up to Approximately 30 months
  ORR is defined as the proportion of participants who had confirmed complete response (CR) or partial response (PR) as determined by investigators per RECIST v1.1.
Phase 1a and Phase 1b: Duration of Response (DOR) as determined by investigators per RECIST v1.1. | Up to Approximately 30 months
  DOR is defined as the time from the first determination of a confirmed objective response until the first documentation of progression or death due to any cause, whichever occurs first.
Phase 1a and Phase 1b: Disease Control Rate (DCR) as determined by investigators per RECIST v1.1. | Up to Approximately 30 months
  DCR is defined as the proportion of participants with best overall response (BOR) of confirmed CR, PR, or stable disease
Phase 1a and Phase 1b: Clinical Benefit Rate (CBR) as determined by investigators per RECIST v1.1. | Up to Approximately 30 months
  CBR is defined as the proportion of participants with BOR of confirmed CR, PR, or stable disease lasting ≥ 24 weeks.
Phase 1b: Progression Free Survival (PFS) as determined by investigators per RECIST v1.1. | Up to Approximately 30 months
  PFS is defined as the time from the date of the first administration of study drug to the date of the first documentation of disease progression or death due to any cause, whichever occurs first.
Phase 1a and Phase 1b: Maximum Serum Concentration (Cmax) of BGB-B167 | Up to Approximately 30 months
Phase 1a and Phase 1b: Minimum Observed Plasma Concentration (Cmin) of BGB-B167 | Up to Approximately 30 months
Phase 1a and Phase 1b: Time to Cmax (Tmax) of BGB-B167 | Up to Approximately 30 months
Phase 1a: Terminal half-life (t1/2) of BGB-B167 | Up to Approximately 30 months
Phase 1a: Area Under the Plasma Concentration-time curve (AUC0-7d) of BGB-B167 | Up to Approximately 30 months
Phase 1a: Clearance (CL) BGB-B167 | Up to Approximately 30 months
Phase 1a: Volume of Distribution at Steady State (Vss) of BGB-B167 | Up to Approximately 30 months
Phase 1a and Phase 1b: Number of Participants with Anti-Drug Antibodies (ADAs) | Up to Approximately 30 months
Phase 1b: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Approximately 30 months